CLINICAL TRIAL: NCT05769998
Title: Development and Improvement of an Acceptance and Commitment-based Treatment for the Prevention of Chronic Pain After Total Knee Arthroplasty
Acronym: NOPAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03M902
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment-based treatment (Experimental): Acceptance and Commitment-based (ACT) treatment including a face-to-face component administered during the patient stay in the rehabilitation unit and an online component including 4 ACT modules with an estimated duration of one month. The treatment is added to the Treatment as Usual provided in the rehabilitation unit.
  Interventions: Behavioral: Acceptance and Commitment-based treatment; Other: Treatment as usual
- Treatment as usual (Other): Usual care including pharmacological therapy and exercise therapy, administered in the rehabilitation unit independently from the project.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment-based treatment — The ACT-based group intervention includes four 1-hour group sessions over two weeks. The treatment manual was developed by the authors of this study following the ACT framework and adapting materials and resources from ACT-based treatments developed for other settings. The focus of the intervention is to provide patients with pain education specific for patients who underwent TKA and to promote psychological flexibility. Each session employs experiential exercises, including mindfulness meditation, and metaphors addressing the core components of ACT.
  Arms: Acceptance and Commitment-based treatment
Other: Treatment as usual — Standard pharmacotherapy and physical exercise plan provided to all the patients in the rehabilitation unit.

SUMMARY:
Reducing the incidence of chronic post-surgical pain after Total Knee Arthroplasty (TKA) is paramount. NOPAIN, a technology-enhanced Acceptance and Commitment-based treatment, will be developed, tested and improved for this purpose. The feasibility of NOPAIN will be evaluated in a small sample of patients listed for TKA at the IRCCS Istituto Auxologico Italiano. Potential pre-surgical and post-surgical predictors of non-response to treatment will be measured and tested using a machine learning algorithm. The results of this study will be employed to improve the content of NOPAIN or for identification of criteria for patient selection. Finally, a randomized controlled clinical trial will be performed. Patients listed for TKA will be randomized to Treatment As Usual (TAU) or to NOPAIN+TAU. Primary outcome will be time to complete pain relief, secondary outcomes will include subjective and objective measurements of quality of life and functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* having an age between 18 and 80 years
* having a diagnosis of OA as determined by medical record review
* having undergone a Total Knee Arthroplasty

Exclusion Criteria:

* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of days for pain disappearance | 6 months
  The first among five consecutive days with pain intensity <3 on a 0-10 Numeric Rating Scale

SECONDARY OUTCOMES:
Presence of chronic pain | 6 months
  WOMAC pain subscale >4
Pain intensity | 6 months
  Pain intensity as measured by a 0-10 Numeric Rating Scale
Knee pain, stiffness and physical function | 6 months
  Subscales of the WOMAC questionnaire
Physical and Mental Quality of Life | 6 months
  Physical and Mental component scores on the SF-12 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Auxologico Mosè Bianchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be uploaded to an online repository
Supporting Information: Study Protocol, SAP
Time Frame: The dataset will be made available upon completion
Access Criteria: The dataset will be uploaded to an online repository